CLINICAL TRIAL: NCT04884893
Title: The Effect of Nitrous Oxide on EEG, a Randomized, Double-blinded Study
Brief Title: Effect of Nitrous Oxide on EEG
Acronym: HUMANOID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R18097M
Record Dates: First submitted 2021-03-09; First posted 2021-05-13 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-03

CONDITIONS: Nitrous Oxide; Electroencephalography; Anesthetic, Inhalation
Keywords: EEG; Slow wave activity; Nitrous oxide; N-methyl-D-aspartate-receptor blockade; Delta wave; Self-reported psychiatric symptoms
MeSH Terms: conditions — Respiratory Aspiration | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent nitrous oxide (Experimental): 10 minutes of 50% nitrous oxide + 10 min 100% oxygen + 10 min 50% nitrous oxide + 10 min 100% oxygen
  Interventions: Drug: Nitrous Oxide
- Continuous nitrous oxide (Experimental): 20 min 50% nitrous oxide + 20 min 100% oxygen
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — 50% nitrous oxide

SUMMARY:
Our recent preclinical observations suggest that monitoring of slow electroencephalogram (EEG) oscillations may be used to predict the efficacy of rapid-acting antidepressants such as ketamine or nitrous oxide. In this project we will carry out critical clinical research on healthy volunteers and study the effects of nitrous oxide on EEG. Results will be used for the design of clinical trials on depressed individuals. The project will be done in collaboration between neuroscientists at the University of Helsinki and clinicians at the Tampere University Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent obtained
2. age between 18 - 40
3. male
4. body mass index 18 - 27

Exclusion Criteria:

1. Age < 18 or > 40
2. Alcohol Use Disorders Identification Test (AUDIT) >6 points
3. Drug Abuse Screening Test 20 (DAST-20) > 0 points
4. Beck Depression Inventory (BDI) > 11 points
5. Symptom Check List 90 (SCL-90) over mean values of Finnish population in any dimensions of the SCL-90 or the global severity index
6. Any respiratory disorder including sleep apnea
7. Any heart illness
8. Epilepsy
9. Known vitamin B12 deficiency

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females excluded due to higher risk of nausea and due to menstrual cycle's effect on EEG
Enrollment: 20 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Slow wave activity | During nitrous oxide administration
  Delta wave in EEG
Slow wave activity | Following 20 minutes after nitrous oxide administration
  Delta wave in EEG

SECONDARY OUTCOMES:
Self-reported psychiatric symptoms | Baseline, 20 minutes after nitrous oxide
  Symptom Check List 90 (SCL-90) is a self-reported questionnaire measuring psychological stress. Results are normed, meaning that test scores can be compared to Finnish reference values. In this study we measure if there is an increase in self-reported psychiatric symptoms after nitrous oxide administration.
Side effects - anxiety | Baseline, 20 minutes after nitrous oxide
  Self reported anxiety on a 0 (no at all) to 5 (very much) scale
Side effects - restlessness | Baseline, 20 minutes after nitrous oxide
  Self reported restlessness on a 0 (no at all) to 5 (very much) scale
Side effects - mood elevation | Baseline, 20 minutes after nitrous oxide
  Self reported mood elevation on a 0 (no at all) to 5 (very much) scale
Side effects - nausea | Baseline, 20 minutes after nitrous oxide
  Self reported nausea on a 0 (no at all) to 5 (very much) scale
Side effects - tension | Baseline, 20 minutes after nitrous oxide
  Self reported tension on a 0 (no at all) to 5 (very much) scale
Side effects - uneasiness | Baseline, 20 minutes after nitrous oxide
  Self reported uneasiness on a 0 (no at all) to 5 (very much) scale
Side effects - tiredness | Baseline, 20 minutes after nitrous oxide
  Self reported tiredness on a 0 (no at all) to 5 (very much) scale
Side effects - numbness | Baseline, 20 minutes after nitrous oxide
  Self reported numbness on a 0 (no at all) to 5 (very much) scale
Side effects - dizziness | Baseline, 20 minutes after nitrous oxide
  Self reported dizziness on a 0 (no at all) to 5 (very much) scale
Side effects - agitation | Baseline, 20 minutes after nitrous oxide
  Self reported agitation on a 0 (no at all) to 5 (very much) scale

CONTACTS AND LOCATIONS:
Overall Officials: Maija-Liisa Kalliomäki, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland